CLINICAL TRIAL: NCT01631539
Title: Chemoembolisation With Irinotecan Loaded DC Bead (DEBIRI) in Combination With Cetuximab and 5FU/LV in the First Line Treatment of Patients With KRAS Wildtype Metastatic Colorectal Cancer (mCRC)
Brief Title: Chemoembolisation With CPT11 Loaded DC Bead With Cetuximab and 5FU/LV in First Line in Patients With KRAS Wildtype mCRC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Eric Van Cutsem, Professor MD PhD Eric Van Cutsem, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-018384-42
Record Dates: First submitted 2011-09-14; First posted 2012-06-29 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Liver Metastases; Colorectal Cancer
Keywords: chemoembolization; DC Bead™; Irinotecan; Cetuximab; 5FU/LV; KRAS; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemoembolization (Other): chemoembolization with DC Bead™ loaded with Irinotecan
  Interventions: Device: DC Bead™; Drug: Cetuximab; Drug: 5 FU; Drug: Irinotecan

INTERVENTIONS:
Device: DC Bead™ — chemoembolization with DC Bead™ loaded with Irinotecan
  Other Names: Irinotecan
Drug: Cetuximab — 400 mg/m² IV at day 1 followed by 250 mg/m² IV weekly
  Other Names: Erbitux
Drug: 5 FU — every 2 weeks IV
  Other Names: 5 fluoro uracyl
Drug: Irinotecan — every 4 weeks chemoembolization

SUMMARY:
The purpose of this study is to assess feasibility of chemoembolization with DC Bead loaded with Irinotecan in combination with Cetuximab and 5FU/LV as a first line treatment for wildtype KRAS unresectable liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
20 patients will be included. The duration of the trial will be approximately 24 months.

Every 8 weeks there will be a tumour lesion assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of stage IV KRAS wild-type colorectal adenocarcinoma, with metastases predominantly in the liver (≥80% of tumor burden) that are deemed unresectable.
2. Primary tumour has been treated with complete surgical resection without evidence of residual tumour
3. Patients must have at least 1 measurable lesion (RECIST criteria)
4. Performance status ECOG 0-1
5. Aged ≥18 years
6. Life expectancy > 3 months
7. No prior chemotherapy for metastatic disease
8. Hematologic function: WBC ≥ 3.0 x 10*9/L, platelets ≥ 100 x10*9/L
9. Adequate organ function as measured by:

   * Serum creatinine £ 1.5 x upper limit of normal (ULN)
   * Serum transaminases (AST & ALT) £ 5 x ULN
   * Bilirubin> 1.5 times the upper limit of the normal range
10. Women of child bearing potential and fertile men are required to use effective contraception (negative βHCG for women of child-bearing age)
11. Signed, written informed consent
12. Patients with patent main portal vein
13. Maximum liver involvement ≤60%

Exclusion Criteria:

1. Presence of CNS metastases
2. Contraindications to FU/LV, Irinotecan or Cetuximab
3. Active bacterial, viral or fungal infection within 72 hours of study entry
4. Women who are pregnant or breast feeding
5. Allergy to contrast media or history of severe hypersensitivity to study drugs.
6. Presence of another concurrent malignancy. Prior malignancy in the last 5 years except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
7. Any contraindication for hepatic embolization procedures:

   * porto-systemic shunt
   * hepatofugal blood flow
   * severe atheromatosis
8. Contraindication to hepatic artery catheterization, such as a patient with severe peripheral vascular disease precluding catheterization
9. Other significant medical or surgical condition, or any medication or treatment regimens, that would place the patient at undue risk, that would preclude the safe use of chemoembolization or would interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of chemoembolization with DC Bead loaded with Irinotecan | after one cycle = after 8 weeks
  Feasibility of the study by measuring the number of enrolled patients who can finish the first cycle of treatment

SECONDARY OUTCOMES:
progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months
  progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Cutsem, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven